CLINICAL TRIAL: NCT04145726
Title: Frailty In Thoracic Surgery for Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mette Siemsen, Doctor of Medical Science, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: H-16020318
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing esophageal resection: All patients undergoing esophageal resection will be included and tested if frail or non-frail. Which means there is no intervention

SUMMARY:
Background: In Demark we se an increasing life expectancy and an increasing incidence of esophageal cancer and gastroesophageal junction (c.esophagus), with an average age of 65 years at diagnosis time. The consequence of this is an increased number of patients in need of esophageal resection. Esophageal cancer is currently treated with chemotherapy, radiotherapy and, whenever possible, esophageal resection. This multimodal treatment has increased survival, but is also associated with significant morbidity, mortality and adverse postoperative quality of life. At present, there is no standardized risk assessment for patients with c.esophagus who have to undergo esophageal resection.

This study evaluates the preoperative risk using the frailty score system, CAF (comprehensive assessment of frailty) score, which identify patients being frail or not based on an assessment of the patient's physical condition.

Purpose: Investigate how many patients that are frail undergoing esophageal resection.

With the assumptions that CAF score can identify frail patients and that frail patients, have an increased risk of postoperative complications. With CAF score, we believe to become better of predicting complications following esophageal resection.

Method: Prospective observational study of patients with c.esophagus undergoing esophageal resection. Plan to include 60 patients over one year period. The patients are deemed frail or not with the use of CAF score, which consist of various smaller physical test and questions.

Postoperativley a follow-up after 30-days, six month and 12 month. At follow-up times, data are collected on the somatic readmissions / diagnoses and vital status. Afterwards we compare complications, mortality and quality of life in frail versus non-frail patients.

Side effects, risks and disadvantages: At present, there is no standardized risk assessment used for preoperative risk assessment for patients with c.esophagus undergoing esophageal resection. The introduction of CAF score, will not expose patients to a risk or side effect, since the course or treatment does not change.

Economy: We consider the study to be economically justified, since we hypothesize that this would lead to fewer readmissions, days of intensive care and shorter hospitalization.

Acquisition: The patients will be 60 years or older and are undergoing esophageal resection. They will receive verbal- and written information preoperatively. At the first appearance they meet our project assistant who will answer any questions. Subsequently, the patients will be asked to sign a consent form.

Publication of test results / research ethics statement: The knowledge and results gained through the research will provide essential scientific information of significans for the future course and treatment of patients undergoing esophageal resection in terms of number of hospital days, intensive days and readmissions.

DETAILED DESCRIPTION:
Background: The incidence of esophageal cancer and gastroesophageal junction (c.esophagus) has increased significantly in recent decades. In addition, an increasing life expectancy is seen in Denmark and the average age for diagnosis of c. Esophagus is 65 years. Consequences of this are that we are currently seeing an increased number of patients in need of esophageal resection. Esophageal cancer is currently treated with chemotherapy and radiotherapy and, whenever possible, esophageal resection. This multimodal treatment has increased survival, but is also associated with significant morbidity, mortality and adverse postoperative quality of life. C. Esophagus is among the top ten causes of cancer-related deaths worldwide.

At present, there is no standardized risk assessment for patients with c.esophagus who have to undergo esophageal resection and the subjective assessment is often poor in predicting the postoperative course. A few studies have examined the objective assessment of patients' biological age, also called "frailty," in patients with esophageal cancer who need to be resected. Frailty is a term used to assess the true biological status of a patient and defined as a patient's impaired resistance to stressors due to a decline in physiologic reserve.

It has been shown that up to 57% of patients are pre-frail and that frailty is associated with high postoperative mortality and morbidity. Therefore, there is a need to validate preoperative frailty assessment in patients with c.esophagus, to find those surgically vulnerable patients who may benefit from pre-habilitation prior to surgery, postoperative or those patients who cannot tolerate surgery at all.

For frailty assessment in surgical patients, several different tools are found in the literature. None of these frailty risk scores are fully validated and therefore widely adopted. In German and Denmark two larger studies investigated frailty with the use of Comprehensive assessment of frailty (CAF) score, in patients undergoing cardiac surgery. They found CAF score to be strong predictor of mortality and morbidity after surgery. CAF score is based on an assessment of the patient's physical condition based on questions about the patient's medical history and daily physical activity as well as performing minor physical tests, consisting of strength, balance and walking speed. If the patient has a poorer physical condition than expected, the patient is deemed frail.

Aim: In an observational prospective study, we will identify and describe the number of frail patients undergoing first time esophageal resection in our department, compare the risk of short-term and long-term complications and compare quality of life in frail versus non-frail patients. Frailty will be assessed with CAF-score.

Hypothesis: Patients deemed frail using the CAF score have increased risk of short-term and long-term complications. With the frailty score we can become better of predicting postoperative complications in patients undergoing esophageal resection.

Method:

A) Patients:

Prospective observational study of patients with c.esophagus undergoing esophageal resection at department of Thoracic Surgery and Abdominal Surgery, Rigshospitalet, University of Copenhagen, Denmark. Expect to include 60 patients over a period of 1 year. With a follow-up of minimum 12 month.

B) Follow-up:

Patients are followed after discharge by searching The Danish National Registry, which contains information an all somatic hospital admissions. From which there will be collected a copy of the patient record for all hospital admissions. Patient records will be assessed for pour predefined outcome measures.

Information about vital status will be achieved by searching the Danish Central Civil Register. The cause of death will be obtained from patients' records and death certificates.

At 30 days postoperatively the patient is seen in the hospital outpatient clinic, where blood samples and quality of life will be performed. After six month and one year we will contact the patients through phone to ask about their quality of life and intake/changes in medicine. The follow-up will be so the first one included is followed until the last one is recruited.

C) The Frailty scoring scale:

Frailty is evaluated by using the comprehensive assessment of frailty (CAF) scoring scale of S. Sündermann (8,10). This is based on a combination of different scoring scales. The first part is based on the Fried criteria: weight loss, self-reported exhaustion, low activity, slowness of gait speed and weakness. Where CAF includes all except weight loss. Self-reported exhaustion are two questions by the original CES-D scale, Center for epidemiological study Depression. Low activity is registered, by asking to instrumental activity of daily living (IADL). The IADL used are, walking, housework, outdoor activity, regular sport and others. Following are kilocalories per week calculated by formula: Kilo Cal= (w x frequency of activity x duration of activity)/2. Slowness, speed in meters per second, where the patient walk 4 meters in normal walking speed and weakness through grip strength by pulling as strong as you can the grasp of the dynamometer in kilograms (kg).

The second part is physical performance tests. Testing the balance, how long you can stand still with your feet together, with one feet halfway in front of the other (semi-tandem) and with one feet completely in front of the other one (tandem). At each position the time is measured and put in to frailty table to score points. In the last element of balance the patients is asked to turn around themselves 360 degrees and again the time is obtained. Then testing the body control, get up and down from a chair three times, put on and remove a jacket and pick up a pen from the floor.

The last part is Laboratory tests including level of serum albumin, Creatinine and calculate Forced expiratory volume in 1 s (FEV1).

At the end two physicians, different from the person observing the CAF test (one cardiac surgeon and one experienced clinician) estimate the patients frailty after the Clinical frailty scale score.

The Clinical frailty scale is from the Canadian Study of Health and Aging, Which is based on a frailty index composed of 70 items, from where you estimate the frailty on a scale 1-7. 1. Very fit: robust, active, energetic, well motivated and fit; these people commonly exercise regularly and are in the most fit group for their age. 2. Well: without active disease, but less fit than people in category 1. 3. Well, with treated comorbid disease: disease symptoms are well controlled compared with those in category 4. 4. Apparently vulnerable: although not frankly dependent, these people commonly complain of being "slowed up" or have disease symptoms. 5. Mildly frail: with limited dependence on others for instrumental activities of daily living. 6. Moderately frail: help is needed with both instrumental and non- instrumental activities of daily living. 7. Severely frail: completely dependent on others for the activities of daily living, or terminally ill.

Finally to get the patients total CAF score, you add each individual test scores together. It has a maximum score of 35 points. That is divided into not frail 1-10, moderately frail 11-25 and severely frail 26-35.

Out from the CAF score, there is an ability to score and use FORECAST (Frailty predicts death One year after elective cardiac surgery test) which include only 5 of CAF items: chair rise, weakness, stair climb, CFS (clinical frailty scale) and Serum creatinine. FORECAST has a maximum score of 14 points, which also is divided into, not frail 0-4, moderately frail 5-7 and severely frail 8-14(10).

Statistics:

Sample size calculation:

Previous study by Chih-Hao Chen et al. (5) have assessed frailty in the cancer esophagus in 61 patients and found a 6-month mortality of 35% in the group of frail patients and 5% in the group of non-frail. The number of frail in this study has been found to be 33% but is seen to be as high as 57%. Based on the above, the following is assumed:

We expect a 6-month mortality of 5% in the non-frail group (P1 = 0.05) We expect a 6-month mortality of 35% in the frail group (P2 = 0.35) We have chosen a significance level of 5% (alpha = 0.05) and power of 80%. At the same time, we expect a distribution of the 1/2 frail group and 1/2 the non-frail group. That is, to achieve the mortality rate described above, we must include at least 30 patients in each group.

Data analysis:

Categorical data will be presented as numbers and percentages and compared using chi square test or Fischer exact test, as appropriate. Continuous data will be described as means with corresponding standard deviations (SD) and compared using students t-test. Time to event for the primary and secondary outcomes will be analyzed using a Cox regression model. Survival curves will be illustrated with Kaplan-Meier plots. A P-value of less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 60 years or older
2. Diagnosed with esophageal cancer being squamous-cell carcinoma or adenocarcinoma
3. Referred to esophageal resection

Exclusion Criteria:

1. Not Danish speaking. Need of an interpreter
2. Severe neuropsychiatric impairment
3. Not cooperative (psychiatric diagnosis)
4. Earlier esophageal resection

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational study of patients with c.esophagus undergoing esophageal resection at department of Thoracic Surgery and Abdominal Surgery, Rigshospitalet, University of Copenhagen, Denmark. Expect to include 60 patients over a period of 1 year. With a follow-up of minimum 12 month.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The portion of frail patients undergoing esophageal resection and 6 -month all-cause of mortality | one year
  Identify number of frail patients undergoing esophageal resection. The patients are deemed frail by score comprehensive assessment of frailty. 6 month all-cause mortality in frail vs. non-frail patients (hospital mortality or death within 6 month postoperatively).

SECONDARY OUTCOMES:
One-year all-cause mortality in frail vs. non-frail patients One-year all-cause mortality in frail vs. non-frail patients One-year all-cause mortality in frail vs. non-frail patients | one year

OTHER OUTCOMES:
postoperatively complications in frail vs. non-frail | one year
  Prolonged ventilation, stroke, extended time of per-operative induced drainage (>8 days), days and readmission in intensive care unit, need for reoperation, wound infection, anastomotic leakage, days on total parenteral nutrition, renal failure until discharged, postoperative Chylus, days of hospitalization, prolonged hospitalization (>14 days), discharged to other hospital or nursing home for ongoing medication or rehabilitation and how many days until discharged to home, registration of The Clavien-Dindo Classification, diabetic status by Hba1c, number of re-hospitalization, estimate the quality of life in frail versus non-frail patients undergoing Esophageal resection. This by using "Functional Assessment of Cancer Therapy-Esophageal"(FACT-E), which is a standard screening system for statement of the patients health condition. Analyze improvement of life quality after surgery in frail vs non-frail

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beckert AK, Huisingh-Scheetz M, Thompson K, Celauro AD, Williams J, Pachwicewicz P, Ferguson MK. Screening for Frailty in Thoracic Surgical Patients. Ann Thorac Surg. 2017 Mar;103(3):956-961. doi: 10.1016/j.athoracsur.2016.08.078. Epub 2016 Oct 6. PMID 27720368
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Allen C, Barber RM, Barregard L, Bhutta ZA, Brenner H, Dicker DJ, Chimed-Orchir O, Dandona R, Dandona L, Fleming T, Forouzanfar MH, Hancock J, Hay RJ, Hunter-Merrill R, Huynh C, Hosgood HD, Johnson CO, Jonas JB, Khubchandani J, Kumar GA, Kutz M, Lan Q, Larson HJ, Liang X, Lim SS, Lopez AD, MacIntyre MF, Marczak L, Marquez N, Mokdad AH, Pinho C, Pourmalek F, Salomon JA, Sanabria JR, Sandar L, Sartorius B, Schwartz SM, Shackelford KA, Shibuya K, Stanaway J, Steiner C, Sun J, Takahashi K, Vollset SE, Vos T, Wagner JA, Wang H, Westerman R, Zeeb H, Zoeckler L, Abd-Allah F, Ahmed MB, Alabed S, Alam NK, Aldhahri SF, Alem G, Alemayohu MA, Ali R, Al-Raddadi R, Amare A, Amoako Y, Artaman A, Asayesh H, Atnafu N, Awasthi A, Saleem HB, Barac A, Bedi N, Bensenor I, Berhane A, Bernabe E, Betsu B, Binagwaho A, Boneya D, Campos-Nonato I, Castaneda-Orjuela C, Catala-Lopez F, Chiang P, Chibueze C, Chitheer A, Choi JY, Cowie B, Damtew S, das Neves J, Dey S, Dharmaratne S, Dhillon P, Ding E, Driscoll T, Ekwueme D, Endries AY, Farvid M, Farzadfar F, Fernandes J, Fischer F, G/Hiwot TT, Gebru A, Gopalani S, Hailu A, Horino M, Horita N, Husseini A, Huybrechts I, Inoue M, Islami F, Jakovljevic M, James S, Javanbakht M, Jee SH, Kasaeian A, Kedir MS, Khader YS, Khang YH, Kim D, Leigh J, Linn S, Lunevicius R, El Razek HMA, Malekzadeh R, Malta DC, Marcenes W, Markos D, Melaku YA, Meles KG, Mendoza W, Mengiste DT, Meretoja TJ, Miller TR, Mohammad KA, Mohammadi A, Mohammed S, Moradi-Lakeh M, Nagel G, Nand D, Le Nguyen Q, Nolte S, Ogbo FA, Oladimeji KE, Oren E, Pa M, Park EK, Pereira DM, Plass D, Qorbani M, Radfar A, Rafay A, Rahman M, Rana SM, Soreide K, Satpathy M, Sawhney M, Sepanlou SG, Shaikh MA, She J, Shiue I, Shore HR, Shrime MG, So S, Soneji S, Stathopoulou V, Stroumpoulis K, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tadese F, Tedla BA, Tessema GA, Thakur JS, Tran BX, Ukwaja KN, Uzochukwu BSC, Vlassov VV, Weiderpass E, Wubshet Terefe M, Yebyo HG, Yimam HH, Yonemoto N, Younis MZ, Yu C, Zaidi Z, Zaki MES, Zenebe ZM, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-years for 32 Cancer Groups, 1990 to 2015: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2017 Apr 1;3(4):524-548. doi: 10.1001/jamaoncol.2016.5688. PMID 27918777
- [Background] Murray P, Whiting P, Hutchinson SP, Ackroyd R, Stoddard CJ, Billings C. Preoperative shuttle walking testing and outcome after oesophagogastrectomy. Br J Anaesth. 2007 Dec;99(6):809-11. doi: 10.1093/bja/aem305. Epub 2007 Oct 24. PMID 17959592
- [Background] Chen CH, Ho-Chang, Huang YZ, Hung TT. Hand-grip strength is a simple and effective outcome predictor in esophageal cancer following esophagectomy with reconstruction: a prospective study. J Cardiothorac Surg. 2011 Aug 15;6:98. doi: 10.1186/1749-8090-6-98. PMID 21843340
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Robinson TN, Eiseman B, Wallace JI, Church SD, McFann KK, Pfister SM, Sharp TJ, Moss M. Redefining geriatric preoperative assessment using frailty, disability and co-morbidity. Ann Surg. 2009 Sep;250(3):449-55. doi: 10.1097/SLA.0b013e3181b45598. PMID 19730176
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Sundermann S, Dademasch A, Praetorius J, Kempfert J, Dewey T, Falk V, Mohr FW, Walther T. Comprehensive assessment of frailty for elderly high-risk patients undergoing cardiac surgery. Eur J Cardiothorac Surg. 2011 Jan;39(1):33-7. doi: 10.1016/j.ejcts.2010.04.013. PMID 20627611
- [Background] Back C, Hornum M, Olsen PS, Moller CH. 30-day mortality in frail patients undergoing cardiac surgery: the results of the frailty in cardiac surgery (FICS) copenhagen study. Scand Cardiovasc J. 2019 Dec;53(6):348-354. doi: 10.1080/14017431.2019.1644366. Epub 2019 Jul 23. PMID 31304801
- [Background] Sundermann S, Dademasch A, Rastan A, Praetorius J, Rodriguez H, Walther T, Mohr FW, Falk V. One-year follow-up of patients undergoing elective cardiac surgery assessed with the Comprehensive Assessment of Frailty test and its simplified form. Interact Cardiovasc Thorac Surg. 2011 Aug;13(2):119-23; discussion 123. doi: 10.1510/icvts.2010.251884. Epub 2011 Mar 4. PMID 21378017